CLINICAL TRIAL: NCT06525753
Title: Weaning is Winning? (WeWin Study): Are Parenteral Nutrition (PN) Graduates Growing Up Healthy?
Brief Title: Weaning is Winning? (WeWin Study)
Status: Recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Erasmus University Medical Center (Erasmus MC) - Sophia Children's Hospital (Unknown)
Responsible Party: Principal Investigator, Jessie Hulst, Staff Physician, The Hospital for Sick Children
Other Study IDs: 1000080824
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-07

CONDITIONS: Intestinal Failure; Parenteral Nutrition
Keywords: Quality of Life; Pediatric
MeSH Terms: conditions — Intestinal Failure; Hyperphagia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SickKids: Patients recruited from the Hospital for Sick Children (SickKids), Toronto, Canada
  Interventions: Other: Weaning off Parenteral Nutrition
- Erasmus: Patients recruited from the Erasmus MC-Sophia Children's Hospital, Rotterdam, the Netherlands
  Interventions: Other: Weaning off Parenteral Nutrition

INTERVENTIONS:
Other: Weaning off Parenteral Nutrition — pediatric intestinal failure patients who have been weaned off parenteral nutrition

SUMMARY:
We propose a multicenter prospective study on pediatric patients with intestinal failure (IF) who weaned off parenteral nutrition (PN).

DETAILED DESCRIPTION:
Children with IF depend on PN. This is associated with frequent and various complications such as metabolic bone disease, micronutrient deficiencies and abnormal body composition. Due to advancements in care, many patients with IF are able to wean off PN; they are so called PN graduates. It is currently not well known how often complications do occur after weaning off PN, and which patients are at highest risk of developing these complications.

ELIGIBILITY:
Inclusion Criteria:

* Parenteral Nutrition graduates for at least 1 year, with a history of intestinal failure.
* Age <18 years at time of inclusion.

Exclusion criteria:

* No consent provided.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Parenteral Nutrition graduates, i.e.: patients weaned off Parenteral Nutrition at time of inclusion for at least 1 year, with a history of intestinal failure, defined as dependence on supplemental PN support for a minimum of 60 days within a 74 consecutive day interval and followed by the Group for Improvement of Intestinal Function and Treatment (GIFT) team (SickKids) or IF team (Erasmus MC) as an outpatient.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2034-06-01 (Estimated)

PRIMARY OUTCOMES:
Complications | From 1 year after weaning off PN to 18 years of age
  Assess the frequency of nutritional complications including poor growth, micronutrient deficiencies, poor bone health, abnormal body composition, and delayed pubertal development in PN graduates.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
All participants will be assigned a unique study ID (identification) known only to the study investigators/coordinators. The unique study IDs will only be identifiable through an encrypted master-linking log stored on a secure hospital server and shared folder that is only accessible to designated study staff on each site.